CLINICAL TRIAL: NCT00484263
Title: The Long Term Effect of Inhaled Hypertonic Saline (6%) in Patients With Non-cystic Fibrosis Bronchiectasis.
Brief Title: The Long Term Effect of Inhaled Hypertonic Saline (6%) in Patients With Non Cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Mrs Caroline Nicolson, The Alfred Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T10716
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: Hypertonic saline 6% -

INTERVENTIONS:
Drug: Hypertonic saline 6% - — Hypertonic saline (6%) - 5mls twice a day via a nebuliser for 12 months

SUMMARY:
The purpose of this study is to determine whether the daily inhalation of nebulised hypertonic saline (6%) will decrease the incidence of pulmonary exacerbations and increase the quality of life for people with non cystic fibrosis bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is a disabling, chronic respiratory condition which significantly impacts on the quality of life of patients who present with chronic sputum production and respiratory infections. The occurrence of pulmonary infections is a strong predictor of morbidity and mortality in this group of people so the primary goal of treatment is to prevent infections caused by the presence of sputum in their lungs.

Physiotherapy is a major aspect of their management and focuses on teaching appropriate airways clearance techniques. Traditionally, the physiotherapy management of sputum retention due to bronchiectasis has included the active cycle of breathing technique which has been demonstrated to enhance airways clearance. For some patients, this treatment is not adequate. The use of nebulised hypertonic saline has been used for patients with cystic fibrosis and has been demonstrated to improve sputum removal and lung function.

The aim of this project is to determine the long term effect of the daily inhalation of hypertonic saline on respiratory infections, quality of life, lung function and hospital admissions in patients with non cystic fibrosis bronchiectasis. Hypertonic saline has been shown to be beneficial as a once only treatment in this patient group, but its' long term effects have not been studied.

Participants will be randomised to two groups - those receiving hypertonic saline (6%) and those receiving isotonic saline (0.9%) - and will be blinded to the treatment that they are receiving. They will be given nebuliser equipment and will be instructed how and when to inhale their medication.

Objective measures will be taken by a blinded assessor before the commencement of the project and then at 3 months, 6 months and 12 months post commencement.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bronchiectasis on high resolution computer tomography
* at least 2 respiratory exacerbations per year over the past 2 years
* producing sputum daily
* in a stable clinical state
* over 18 years of age.

Exclusion Criteria:

* cystic fibrosis
* Positive response to hypertonic saline challenge - FEV 1 decreased by ≥ 15%
* FEV 1 ≤ 1L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of pulmonary exacerbations | One year

SECONDARY OUTCOMES:
- St George Respiratory questionnaire - Leicester Cough Questionnaire - Lung Function Tests | One year

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holland, PhD, BAppSc, Study Chair — The Alfred; Caroline H Nicolson, MPhysio, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, Belousova EG, Xuan W, Bye PT; National Hypertonic Saline in Cystic Fibrosis (NHSCF) Study Group. A controlled trial of long-term inhaled hypertonic saline in patients with cystic fibrosis. N Engl J Med. 2006 Jan 19;354(3):229-40. doi: 10.1056/NEJMoa043900. PMID 16421364
- [Background] Kellett F, Redfern J, Niven RM. Evaluation of nebulised hypertonic saline (7%) as an adjunct to physiotherapy in patients with stable bronchiectasis. Respir Med. 2005 Jan;99(1):27-31. doi: 10.1016/j.rmed.2004.05.006. PMID 15672845
- [Derived] Nicolson CH, Stirling RG, Borg BM, Button BM, Wilson JW, Holland AE. The long term effect of inhaled hypertonic saline 6% in non-cystic fibrosis bronchiectasis. Respir Med. 2012 May;106(5):661-7. doi: 10.1016/j.rmed.2011.12.021. Epub 2012 Feb 19. PMID 22349069